CLINICAL TRIAL: NCT04000802
Title: Prospective Evaluation of the Decision-making During Multidisciplinary Meetings for Digestive Cancers
Brief Title: Evaluation of the Decision-making During Multidisciplinary Meetings for Digestive Cancers
Status: Completed | Type: Observational
Sponsor: Moroccan Society of Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: MODE_INO
Record Dates: First submitted 2019-06-22; First posted 2019-06-27 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Decision Making; Quality of Health Care; Neoplasms/Therapy; Patient Care Team
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: response to questionnary — No intervention. Observational study

SUMMARY:
Nowadays, the recommended approach for decision-making for oncology patients is based on multidisciplinary meetings (MDT). However, the quality of decision-making during MDT depends on other factors such as the quality of presentation of clinical cases, the degree of participation of different specialists.

In this study, the investigators will evaluate the decision-making during digestive oncology MDT using the validated "Metric Of Decision-Making" tool (MDT-MODe), in the national institute of oncology (Rabat, Morocco).

DETAILED DESCRIPTION:
Multidisciplinary cancer meetings are a multidisciplinary discussion and decision-making process for a patient with cancer. It allows a sharing of knowledge and decision-making, taking into account the opinion of all the specialists involved in the treatment of cancer, in order to propose the best possible decision for the patient. Nevertheless, the quality of decision-making during CPR depends on other factors such as the quality of presentation of clinical cases, the degree of participation of different specialists and the dynamics of meetings.

There are several validated tools for the quantitative assessment of the decision-making mode during CPRs. The best known is the Metric Of Decision-Making (MDT-MODe). MDT-MODe is a validated tool for the observational evaluation of teamwork and the quality of decision-making during cancer CPR.

MDT-MODe is designed to encourage teams to make holistic decisions tailored to each patient and allows an observer to assess, on a case-by-case basis, in a quantitative and objective way:

The quality of the clinical information (antecedents, radiological pathologies, pathological, comorbid, psychosocial problems and patients' points of view) Contribution to decision-making in teams of key professional groups (surgeons, physicians, oncologists, nurses, health professionals, radiologists, pathologists) Taken together, these notes provide an indication of the quality of team decision-making.

In this study, the investigators will evaluate the decision-making during digestive oncology MDT using the validated "Metric Of Decision-Making" tool (MDT-MODe), in the national institute of oncology (Rabat, Morocco).

ELIGIBILITY:
Inclusion Criteria:

* All consecutive cases presented during multidisciplinary cancer meeting for digestive cancer.

Exclusion Criteria:

* Cases not registered in the electronic health record system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Observations were carried out at digestive oncology multidisciplinary meetings at The National Institute of Oncology in Rabat, Morocco. The meetings are held once a week.
  The study will be performed between the 23rd of May and the 4th of July 2019.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
MODE-MDT scores | 60 days from the multidisciplinary team meeting
  The scores of the Metric Of Decision-Making tool during multidisciplinary team meeting for digestive cancer. The instrument include 10 questions rated from 1 to 5. Higher scores indicate better results. The instrument include questions about the quality of clinical information (History, radiological, pathological, comorbid health conditions, psychosocial issues, and patients' views) and the contribution to team decision making of key professional groups (Surgeons, physicians, oncologists, nurses, allied healthcare professionals, radiologists, pathologists and MDT coordinators) ans a question about the decision (Clear, deferred, no decision. Each question is analyzed separately (mean, median, standard deviation, quartiles).

SECONDARY OUTCOMES:
Decision reached | 60 days from the multidisciplinary team meeting
  The rate of cases with decisions during multidisciplinary team meetings (Clear decision about treatment in the MODE-MDT instrument).
Decision factors | 60 days from the multidisciplinary team meeting
  Predictive factors for reaching a clear decision about treatment during multidisciplinary team meetings. The factors analyzed are the question of the MODE-MDT instrument.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institut of oncology, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: No